CLINICAL TRIAL: NCT06302881
Title: One Novel Transfer Learning-based CLIP Model Combined With Self-attention Mechanism for Differentiating the Tumor-stroma Ratio in Pancreatic Ductal Adenocarcinoma: a Multi-center Retrospective Cohort Study
Brief Title: Differentiating Tumor-stroma Ratio in Pancreatic Ductal Adenocarcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Liao Hongfan, principal investigator, department of radiology,the first affiliated hospital of chongqing medical university, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: liaohongfan
Record Dates: First submitted 2024-02-29; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic ductal adenocarcinoma; Tumor stroma ratio; Contrastive language-image pretraining; Self-attention mechanism; Multi-modality feature fusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- low TSR and high TSR group: The assessment of the tumor-stroma ratio (TSR) entailed measuring the percentage of tumor and stroma constituents. Based on earlier research, 5/5 was deemed as ideal threshold of TSR measurement.

SUMMARY:
This study introduces a novel transfer learning-based contrastive language-image pretraining adapter (CLIP-adapter) model for predicting the tumor-stroma ratio (TSR) in pancreatic ductal adenocarcinoma (PDAC) using preoperative dual-phase CT images. The primary aim is to develop an efficient and accessible tool for risk stratification and personalized treatment planning.

DETAILED DESCRIPTION:
The proposed novel Contrastive Language-Image Pretraining-Adapter (CLIP-adapter) model, leveraging transfer learning, framing CLIP and a self-attention mechanism for predicting TSR in PDAC, in order to exhibit high performance in distinguishing low and high TSR PDAC in the test cohort. We speculated the CLIP-adapter model outperformed single-phase models, specifically CLIP models based on arterial or venous phase images alone. The addition of a feature fusion module could enhance the model's differentiation capacity, emphasizing its superiority over single-phase models. Besides, the model we designed utilized both image and text information during network training, instead of focusing on images only. This underscores the importance of comprehensive assessment in PDAC imaging evaluation, with the potential to contribute to risk stratification and personalized treatment planning.

ELIGIBILITY:
Inclusion Criteria:

1. patients with pathologically proven PDAC by surgical resection
2. patients who underwent CT scan within a month before surgery
3. observable pancreatic lesions on available images.

Exclusion Criteria:

1. any anti-cancer therapy before CT scanning
2. conspicuous interference or significant motion distortions found on images
3. partial clinical data
4. patients with liver metastases or peritoneal carcinomatosis prior to surgical intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 207 patients were chosen from three independent4 hospitals: the First Affiliated Hospital of Chongqing Medical University (FAHCQMU), Daping Hospital of Army Medical University (DPHAMU), and the Third Affiliated Hospital of Chongqing Medical University (TAHCQMU).
Sampling Method: Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
The diagnostic AUC value of pancreatic ductal adenocarcinoma with deep learning algorithm. | 1 year
  AUC=(Sensitivity+Specificity)-1

SECONDARY OUTCOMES:
The diagnostic accuracy of pancreatic ductal adenocarcinoma with deep learning algorithm. | 1 year
  The diagnostic accuracy of pancreatic ductal adenocarcinoma with deep learning algorithm.
The diagnostic sensitivity of pancreatic ductal adenocarcinoma with deep learning algorithm. | 1 year
  The diagnostic sensitivity of pancreatic ductal adenocarcinoma with deep learning algorithm.
The diagnostic specificity of pancreatic ductal adenocarcinoma with deep learning algorithm. | 1 year
  The diagnostic specificity of pancreatic ductal adenocarcinoma with deep learning algorithm.
The diagnostic positive predictive value of pancreatic ductal adenocarcinoma with deep learning algorithm. | 1 year
  The diagnostic positive predictive value of pancreatic ductal adenocarcinoma with deep learning algorithm.
The diagnostic negative predictive value of pancreatic ductal adenocarcinoma with deep learning algorithm. | 1 year
  The diagnostic negative predictive value of pancreatic ductal adenocarcinoma with deep learning algorithm.

IPD SHARING:
Plan to Share IPD: Undecided